CLINICAL TRIAL: NCT06248749
Title: The Effect Of Intravenous Iron In Treating Anemia In Ovarian Cancer Patients In Saskatchewan: A Phase-III, Open-Label, Randomized Trial (IIOVS-01)
Brief Title: Effect of Intravenously Iron Infusion on the Prevention and Treatment of Anemia in Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Maryam Al-Hayki, Gyn Oncologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIOVS-01
Record Dates: First submitted 2023-01-27; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Anaemia in Ovarian Carcinoma
MeSH Terms: interventions — ferryl iron; iron isomaltoside 1000; ferric derisomaltose; ferric gluconate; Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective, randomized [1:1] controlled, Phase III study of Iron Sucrose, Iron Gluconate or Iron Isomaltoside (Treatment group A) versus No Iron Infusion treatment (Control group B) in participants diagnosed with ovarian cancer and with iron deficiency anemia. The primary objective of the study is to assess the efficacy of iron infusion, as measured by the primary endpoint, of Group A versus Group B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Infusion Arm (Experimental): Group A: Treatment study group All patients will be treated with iron infusion for Hgb lower than 100 g/L and/or TSAT < 20%.
  Interventions: Drug: IV iron
- No Iron Infusion (No Intervention): Group B: No iron Infusion

INTERVENTIONS:
Drug: IV iron — Intravenous Iron supplement
  Other Names: iron isomaltoside (Monofer, Monoferric) ferric gluconate (FG) iron sucrose (IS)
  Arms: Iron Infusion Arm

SUMMARY:
Cancer related anemia (CRA) is a common sign occurring in more than 30% of patients at diagnosis, prior to initiation of antineoplastic therapy. Anemia is known to impact survival, disease progression, treatment efficacy, and the patient's quality of life.

Proinflammatory cytokines, mainly IL-6, which are released by both tumor and immune cells, play a pivotal action in CRA etiopathogenesis: they promote alterations in erythroid progenitor proliferation, erythropoietin (EPO) production, survival of circulating erythrocytes, iron balance, redox status, and energy metabolism, all of which can lead to anemia. Chronic inflammatory conditions such as cancer influences a compromised nutritional status, which in-turn may contribute to anemia.

This study aims to study the role of intravenous (IV) iron infusion in the management of anemia presented in patients previously treated or currently being treated for ovarian cancer. The study aims to identify the safety and efficacy of IV iron infusion on anemia in ovarian cancer patients, and the effect on quality of life and overall survival

DETAILED DESCRIPTION:
This is an open label, prospective, randomized [1:1] controlled, Phase III study of Iron Sucrose, Iron Gluconate or Iron Isomaltoside (Treatment group A) versus No Iron Infusion treatment (Control group B) in participants diagnosed with ovarian cancer and with iron deficiency anemia. The primary objective of the study is to assess the efficacy of iron infusion, as measured by the primary endpoint, of Group A versus Group B.

The study treatment is divided into two groups (Arms):

Group A: Treatment study group

All patients will be treated with iron infusion for Hgb lower than 100 g/L and/or TSAT < 20%. Blood transfusion may also be given based on physician's discretion whenever indicated:

1. When Hgb level is < 70 g/L or in case of emergency and/or rapid blood loss.
2. Blood transfusion may be given to keep active treatment (chemotherapy, surgery, PARP inhibitors, hormonal, radiation) intervals as scheduled and not to exceed the maximum 4 weeks.
3. Based on current practice and NCCN guidelines, co-investigators/treating physicians are encouraged to avoid giving blood transfusion for Hgb >70g/L, provided the patient is stable and asymptomatic.
4. Blood transfusion can be combined with iron infusion.
5. Blood transfusion can be given when indicated if there is lack of response to iron infusion. Expected iron infusion response is expected at 8 weeks or less after treatment (from the preceding dose of a single IV iron order/treatment). For example, Isomatoside, monoferric is given as one dose, where iron gluconate is fractionated over 6 doses and iron sucrose is fractionated into 3 doses.

Group B: Control group

1. May receive blood transfusion when Hgb level is <70 g/L or in case of emergency and/or rapid blood loss.
2. Based on current practice and NCCN guidelines, co-investigators/treating physicians are encouraged to avoid giving blood transfusion for Hgb >70 g/L, provided the patient is stable and asymptomatic.
3. The decision to give blood transfusion for Hgb >70 g/L shall be based on the treating physician's discretion:

   1. symptomatic patient
   2. to maintain active treatment schedule
   3. to prepare the patient for surgery or an interventional procedure

ELIGIBILITY:
INCLUSION CRITERIA:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Age and Sex: Female participants aged 18 years or more (>/=18 years) at the time of informed consent.
2. Type of Participant: Participants who are willing and able to comply with all scheduled visits, laboratory tests, lifestyle considerations, treatment plan, and any other study procedures.
3. Disease Characteristics: Histologically confirmed primary epithelial invasive ovarian cancer of any grade, including serous, mucinous, endometrioid, clear cell, transitional, squamous and carcinosarcoma. Cancer must be FIGO stage IC-IV.
4. Presence of measurable disease per RECIST v1.1, as assessed by investigator and evidenced by available baseline tumor scan. At least 1 target lesion of 10mm.

   Note: Baseline Scan is defined as the last scan prior to the date of randomization.
5. Patients should be eligible for active cancer treatment ECOG less or equal to 2 and life expectancy must be more than 6 months.
6. Received no more than two (2) systemic lines of chemotherapy (to allow for a ~3 years follow up).
7. Patients on any active cancer treatment or with history of previous chemotherapy, surgery, radiation, PARP (Poly-ADP Ribose polymerase), biologics and hormonal treatment.
8. Patients on neoadjuvant, adjuvant, advanced cancer treatment.
9. Perioperative patients having upfront surgery (can be randomized after frozen section) or at interval or secondary debulking surgery.
10. Informed Consent: Capable of giving signed informed consent.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Patients would not consent for IV iron infusion or blood transfusion (Example: Jehovah's Witness).
2. History of known severe hypersensitivity to IV iron transfusion with the study iron products.
3. Medical conditions with contraindication to IV iron infusion or blood transfusion (Example:

   iron overload, hemosiderosis, decompensated liver cirrhosis or active hepatitis.)
4. Palliative patients with life expectancy 6 months or less.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biological female
Enrollment: 200 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Hgb>100g/L (Hemoglobin) | every 3 weeks during treatment, then every 3 months during follow-up, up to 3 years.
  by ongoing monitoring of patient Hgb status for patients on active treatment every 3 weeks and patients in follow-up every 3 months. Effect of Iron infusion on response to chemotherapy.
Safety of IV iron | At every visit through study completion, up to 3 years.
  Measure the safety of IV iron including type and frequency of AEs, SAEs, TEAEs, discontinuation due to AEs and outcome of AE treatment. It will be compared to AEs (including frequency, SAEs, TEAs, discontinuation due to AEs and outcome of AEs treatment) of blood transfusion and it will be compared to literature data on IV iron.
Efficiency of IV iron | every 3 weeks during treatment, then every 3 months during follow-up, up to 3 years.
  To assess the efficiency of IV iron, Hgb will be frequently assessed as per the study protocol. Hgb will be compared to baseline level, looking at substantial increase of Hgb of about 20 g/L increase within maximum 8 weeks (study estimated response time).
Time to response | Hgb will be checked just prior to treatment and then biweekly until week 8 or whenever Hgb rises at least by 20 g/L through the treatment period, upto 3 years.
  Time to response will be measured in every patient treated with IV iron from the time of treatment until substantial increase in Hgb from baseline 20 g/L. Hgb will be checked just prior to IV iron and then biweekly until week 8 or whenever Hgb rises at least by 20 g/L
Delay In Chemotherapy | Throughout study completion, up to 3 years.
  Timing of chemotherapy will be recorded and that will be compared to the standard treatment protocol. Any delay of chemotherapy schedule due to "anemia" will be flagged and recorded in all participants. These data will be compared between the two study groups.
Change in QOL (quality of Life) | At screening, then Post treatment (every 6 months) up to 3 years.
  To measure any change from baseline QOL of both study groups and compare the difference of QOL in Group A (the group receiving IV infusion to correct anemia) compared to Group B. This will be done by comparing scores on the QOL questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Al-Hayki, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No